CLINICAL TRIAL: NCT01072019
Title: Comparative Clinical Study of the Vanguard® Knee System Using Signature™ Custom Guides & Conventional Techniques
Brief Title: A Randomized Prospective Trial of Total Knee Arthroplasty Options Comparing Standard Knee Cutting Guides and MRI Generated Patient Specific Custom Cutting Guides
Acronym: Cutting Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0018; Ortho.CR.K018.10 (Other: Biomet)
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard knee cutting guides (Active Comparator): Standard cutting guides use traditional instrumentation to determine knee implant positions. During surgery, a rod is placed in the leg bone and the cutting guide is attached to that rod.
  Interventions: Other: Instrument
- MRI generated patient specific custom cutting guides (Active Comparator): Patient specific cutting guides are custom-made for each patient based on Magnetic Resonance Imaging (MRI). Before surgery, MRI of the knee is done and used to create a cutting guide that is formed to the exact shape of the knee. The patient specific cutting guides have platforms that can be attached to the bone, so the rod does not need to be placed in the leg bone.
  Interventions: Other: Instrument

INTERVENTIONS:
Other: Instrument — Randomization to instrumentation to be used for primary total knee replacement; either standard knee cutting guides or MRI generated patient specific custom cutting guides.
  Other Names: Vanguard® Knee System; Signature™ Custom Guides

SUMMARY:
The purpose of this study is to determine the surgical and clinical outcomes of patients receiving total knee replacement with the same implant using two different types of cutting guides during surgery:

1. Standard knee cutting guides;
2. MRI generated patient specific custom cutting guides.

Both types of cutting guides used in this study are registered with the U.S. Food and Drug Administration (FDA) and are routinely used for knee replacement surgery. However, it is unknown if one type of cutting guide has risks or benefits over the other.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75
* Diagnosis of osteoarthritis of the knee and qualify for surgery, as indicated by one of the following:
* Painful and disabled knee joint resulting from osteoarthritis where one or more compartments are involved;
* Correction of varus or valgus.
* Willing to participate and return for follow-up study visits.

Exclusion Criteria:

* Infection
* Sepsis
* Osteomyelitis
* Uncooperative patient or patient with neurologic disorders who is incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction
* Marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency
* Muscular atrophy
* Neuromuscular disease
* Incomplete or deficient soft tissue surrounding the knee
* Previous osteotomy
* Diagnosis of rheumatoid arthritis
* Previous patella fracture or surgery
* Previous healed tibia or femur fractures
* Previous joint replacement surgery
* Cannot have an MRI
* Patients receiving single-stage bilateral total knee arthroplasty (TKA)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Patient dissatisfaction following primary total knee replacement. | Preoperatively, intraoperatively, and at four to six weeks, three months, six months, and one year postoperatively.

SECONDARY OUTCOMES:
Postoperative recovery time following primary total knee replacement. | Immediate postoperative period (prior to discharge) and at four to six weeks, three months, six months, and one year postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan M Nunley, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States